CLINICAL TRIAL: NCT03720314
Title: Microbiota and Metabolite Profiles Linked to Severity in Irritable Bowel Syndrome
Brief Title: Microbiota Profiling in IBS
Acronym: IBSQUtrition
Status: Completed | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government); Ingredia S.A. (Industry); Nexira (Industry); Naturex (Other); Bioiberica (Industry); Wecare (Other); Roquette Freres (Industry); Darling (Unknown); Winclove Bio Industries BV (Industry)
Responsible Party: Sponsor
Other Study IDs: NL64950.081.18
Record Dates: First submitted 2018-08-06; First posted 2018-10-25 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2018-11

CONDITIONS: Irritable Bowel Syndrome; Microbial Colonization; Dietary Habits
MeSH Terms: conditions — Irritable Bowel Syndrome; Communicable Diseases; Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will hand in fecal samples for microbiota composition analysis, which will be done using 16r RNA technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBS: Irritable bowel syndrome patients
  Interventions: Other: NA observational study
- control: healthy controls
  Interventions: Other: NA observational study

INTERVENTIONS:
Other: NA observational study — observational study

SUMMARY:
This study investigates differences in microbiota profiles and metabolite levels between mild and severe IBS patients, compared to matched healthy controls. Two fecal samples, with one month in between, will be analyzed. Secondary parameters such as dietary intake, quality of life and stool pattern will be assessed.

DETAILED DESCRIPTION:
Rationale: Irritable Bowel Syndrome (IBS) is a gastro-intestinal disorder that strongly affects Quality of Life and impairs daily functioning. However, the aetiology and pathophysiology has been poorly understood. Studies suggest that intestinal microbiota in IBS is altered, however a general consensus remains elusive. This may be due to the large individual variation in microbiota and IBS symptoms, and the cross-sectional designs. Moreover, other factors like diet, wellbeing and metabolite profiles are often not taken into account. New evidence is suggesting that IBS severity may be an important factor in microbiota composition.

Objective: To determine faecal microbiota composition and metabolite production (such as acetate, propionate and butyrate), and investigate differences between healthy controls and mild or severe patients IBS. Moreover, to investigate whether (clinical) parameters such as symptom severity fluctuated, and if these fluctuations are associated with an alteration in faecal microbiota composition and metabolite production, one month after baseline, compared to healthy controls.

Study design: This study is a repeated cross-sectional study, with two data collection points (baseline, and after one month).

Study population: For this study, 100 IBS patients and 30 healthy controls will be recruited. After the first data collection point (T1), the 30 most mild and 30 most severe IBS patients will be included for data collection at T2 (after one month). All participants will be aged between 18 and 65 years.

Intervention (if applicable): Not applicable. Main study parameters/endpoints: primary endpoint of this study is microbiota composition and metabolite profiles, and the difference between groups and possible change after one month. These are assessed two faecal samples, which are analysed by 16S rRNA gene-based microbiota profiling. Secondary parameters are dietary intake, Quality of Life, depression and anxiety scores, and stool consistency and frequency, which are assessed by validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* IBS patients that meet the Rome IV criteria, or healthy subjects with no gastro-intesitnal complaints
* In close proximity of Wageningen (max. 50 km)
* Signed informed consent.
* After baseline measurements, IBS severity will be checked using the IBS-SSS. Participants will be included for follow-up one month later, when they have the most mild symptoms (n=30) or most severe (n=30) symptoms.

Exclusion Criteria:

* Presence of gastro-intestinal diseases, such as celiac disease, Crohn's disease, or Ulcerative colitis.
* Have a history of intestinal surgery that might interfere with study outcomes. This does not include an appendectomy or cholecystectomy.
* Presence of significant systemic diseases, such as diabetes mellitus, cancer, cardiovascular disease or respiratory disease.
* Female participants: currently pregnant or breast-feeding.
* Use of antibiotic treatment less than 3 months before start of the study and no use of antibiotics during the study.
* You are participant in another study during this study.
* Are an employee or student of the Division of Human Nutrition, Food and Biobased Research or Laboratory of Microbiology, of Wageningen University & Research.
* Unwilling or unable to fulfil study criteria.
* If they are not selected in the most mild or most severe group after T1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 IBS patients, and 30 healthy matched controls. After baseline measurements, the 30 most mild IBS and 30 most severe IBS will be follow-up one month later. n=40 IBS drops out after baseline. Healthy controls will be matched with mild IBS patients, based on age, gender and BMI.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Change in microbiota composition | baseline, and one month later
  microbiota composition will be measured in fecal samples, using 16S rRNA technique
Change in Short chain fatty acid levels | baseline, and one month later
  Metabolite levels will be measured in fecal samples, using HPLC method

SECONDARY OUTCOMES:
Dietary intake | baseline
  Habitual dietary intake and habits will be measured using a Food Frequency Questionnaire.
Change in Stool pattern | baseline, and one month later
  Using the bristol stool chart, and questions on frequency
Change in Gastro-intestinal complaints | baseline, and one month later
  will be measured using the validated questionnaire IBS-Symptom Severy Score (IBS-SSS). These results range from 0 - 500, and defines subjects in categories. <75 will be considered control/remission, 75-175 is considered mild complaints, 175-300 is considered moderate complaints, >300 is considered severe complaints. Based on results at baseline, the IBS group will be split into most mild and most severe IBS subjects.
Change in Anxiety and Depression screening scores | baseline, and one month later
  Using the questionnaire Hospital Anxiety and Depression Scale (HADS). Seperate scores for anxiety and depression will be calculated, ranging from 0 to 21. Subjects can be considered a "case" of depression and anxiety if scores are above 8.
Change in Quality of Life scores | baseline, and one month later
  The questionnaire IBS-Quality of life (IBS-QoL) will be administered, which calculates a score, ranging from 0 - 100. A higher score indicates a good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Witteman, Prof MD PhD, Principal Investigator — Wageningen University & Research
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data will be processed anonymously. Results will be shared in peer reviewed publications

REFERENCES:
- [Derived] Wang T, van Dijk L, Rijnaarts I, Hermes GDA, de Roos NM, Witteman BJM, de Wit NJW, Govers C, Smidt H, Zoetendal EG. Methanogen Levels Are Significantly Associated with Fecal Microbiota Composition and Alpha Diversity in Healthy Adults and Irritable Bowel Syndrome Patients. Microbiol Spectr. 2022 Dec 21;10(6):e0165322. doi: 10.1128/spectrum.01653-22. Epub 2022 Nov 2. PMID 36321894

DOCUMENTS (1):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT03720314/Prot_000.pdf